CLINICAL TRIAL: NCT00968149
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Comparing Montelukast With Placebo in Pediatric Patients Age 2 Through 14 Years With Seasonal Allergic Rhinitis
Brief Title: A Study Comparing Montelukast With Placebo in Children With Seasonal Allergic Rhinitis (0476-219)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-219; MK0476-219; 2009_652
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2009-12-11 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: montelukast sodium
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — one montelukast chewable tablet daily at bed time for 2 weeks, 4 mg for patients aged 2-5 years and 5 mg for patients 6-14 years
  Arms: 1
Drug: Comparator: Placebo — one placebo chewable tablet daily at bed time for 2 weeks
  Arms: 2

SUMMARY:
This study will evaluate the effect of montelukast compared to placebo in children during the spring allergic rhinitis season.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of allergic rhinitis symptoms which flare up during the study season
* Patient is a non-smoker
* Patient is in otherwise good health
* Patient is able to chew a tablet

Exclusion Criteria:

* Patient is hospitalized
* Patient is pregnant or nursing mother, or <8 weeks post partum
* Patient and/or parent intend to move or vacation away from home during the trial
* Patient has had a major surgical procedure within 4 weeks of the prestudy visit
* Patient has been treated in an emergency room or hospitalized for asthma within 3 months prior to study
* Patient has an upper respiratory, eye, or sinus infection, or a history of any of these within 3 weeks prior to study
* Patient has a recent history of a psychiatric disorder or attention deficit hyperactivity disorder

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 413 (Actual)
Dates: Start 2001-03; Primary Completion 2001-06 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bisgaard H, Skoner D, Boza ML, Tozzi CA, Newcomb K, Reiss TF, Knorr B, Noonan G. Safety and tolerability of montelukast in placebo-controlled pediatric studies and their open-label extensions. Pediatr Pulmonol. 2009 Jun;44(6):568-79. doi: 10.1002/ppul.21018. PMID 19449366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty one study sites in the United States.
  Prime Therapy Period: Mar-2001 to Jun-2001.
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime rhinitis symptoms score during the run-in period were excluded from randomization.
Groups:
- Montelukast 4 mg and 5 mg: Patients aged 2 to 5 years: montelukast 4 mg chewable tablet orally once daily at bedtime for 2 weeks. Patients aged 6 to 14 years: montelukast 5 mg chewable tablet orally once daily at bedtime for 2 weeks.
- Placebo: Patients aged 2 to 5 years: montelukast 4 mg matching-image placebo chewable tablet orally once daily at bedtime for 2 weeks. Patients aged 6 to 14 years: montelukast 5 mg matching-image placebo chewable tablet orally once daily at bedtime for 2 weeks.
Period: Overall Study
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Started | 280 | 133
Completed | 269 | 127
Not Completed | 11 | 6
Not completed — Adverse Event | 5 | 1
Not completed — Lack of Efficacy | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 4 mg and 5 mg | Placebo | Total
Number analyzed (Participants) | 280 | 133 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (3.7) | 8.4 (3.8) | 8.0 (3.7)
Sex/Gender, Customized [Number; unit: participants]
  Boys | 157 | 77 | 234
  Girls | 123 | 56 | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs)
Description: A clinical adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 2 weeks
Population: All patients who took study medication during the 2-week, double-blind treatment period were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 280 | 133
Participants
  With CAEs | 73 | 35
  Without CAEs | 207 | 98

2. Secondary Outcome: Number of Patients With Serious CAEs
Description: Serious CAEs are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 2 weeks
Population: All patients who took study medication during the 2-week, double-blind treatment period were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 280 | 133
Participants
  With Serious CAEs | 1 | 0
  Without Serious CAEs | 279 | 133

3. Secondary Outcome: Number of Patients With Drug-related CAEs
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) CAEs
Time Frame: 2 weeks
Population: All patients who took study medication during the 2-week, double-blind treatment period were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 280 | 133
Participants
  With Drug-related CAEs | 10 | 5
  Without Drug-related CAEs | 270 | 128

4. Secondary Outcome: Number of Patients Who Were Discontinued Due to CAEs
Time Frame: 2 weeks
Population: All patients who took study medication during the 2-week, double-blind treatment period were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 280 | 133
Participants
  Discontinued Due to CAEs | 5 | 1
  Did Not Discontinue Due to CAEs | 275 | 132

5. Secondary Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs)
Description: A laboratory adverse experience (LAE) is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: 2 weeks
Population: All patients who took study medication during the 2-week, double-blind treatment period and had at least one laboratory test post baseline were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 272 | 129
Participants
  With LAEs | 2 | 3
  Without LAEs | 270 | 126

6. Secondary Outcome: Number of Patients With Serious LAEs
Description: Serious LAEs are any LAEs occurring at any dose that: Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 272 | 129
Participants
  With Serious LAEs | 0 | 0
  Without Serious LAEs | 272 | 129

7. Secondary Outcome: Number of Patients With Drug-related LAEs
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 272 | 129
Participants
  With Drug-related LAEs | 1 | 2
  Without Drug-related LAEs | 271 | 127

8. Secondary Outcome: Number of Patients Who Were Discontinued Due to LAEs
Time Frame: 2 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Number analyzed (Participants) | 272 | 129
Participants
  Discontinued Due to LAEs | 0 | 0
  Did Not Discontinue Due to LAEs | 272 | 129

ADVERSE EVENTS:
Time Frame: During the 2-week, double-blind treatment period
Description: Patients were monitored for adverse experiences During the 2-week, double-blind treatment period; no adverse experience was suggested. Adverse experiences were recorded at each clinic visit on the Adverse Experience Case Report Forms
Arm/Group | Montelukast 4 mg and 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/280 | 0/133
Other Adverse Events (participants affected / at risk) | 73/280 | 35/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast 4 mg and 5 mg (N=280) | Placebo (N=133)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Montelukast 4 mg and 5 mg (N=280) | Placebo (N=133)
Abdominal Pain (General disorders) | 4 | 2
Asthenia/Fatigue (General disorders) | 2 | 0
Body Ache (General disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Enuresis (General disorders) | 0 | 1
Facial Edema (General disorders) | 1 | 0
Fever (General disorders) | 7 | 4
Purulent Discharge (General disorders) | 1 | 1
Upper Respiratory Infection (Infections and infestations) | 6 | 2
Viral Infection (Infections and infestations) | 1 | 1
Viral Syndrome (Infections and infestations) | 2 | 0
Ecchymosis (Cardiac disorders) | 2 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 4 | 5
Allergic Conjunctivitis (Eye disorders) | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Conjunctival Edema (Eye disorders) | 1 | 0
Conjunctival Injection (Eye disorders) | 2 | 1
Epistaxis (Vascular disorders) | 4 | 4
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal Turbinate Abnormality (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ophthalmic Infection (Eye disorders) | 1 | 0
Otic Pain (General disorders) | 1 | 1
Otitis (Ear and labyrinth disorders) | 1 | 1
Otitis Externa (Ear and labyrinth disorders) | 1 | 0
Otitis Media (Ear and labyrinth disorders) | 6 | 2
Pharyngitis (General disorders) | 9 | 2
Sinusitis (General disorders) | 3 | 0
Tonsillar Disorder (General disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Dream Abnormality (Nervous system disorders) | 3 | 1
Head Trauma (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 2
Hyperkinesia (Nervous system disorders) | 1 | 1
Insomnia (Nervous system disorders) | 1 | 1
Sleep Disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Behavioral Disturbance (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczematous Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Excoriation (Skin and subcutaneous tissue disorders) | 1 | 0
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Venomous Bite/Sting (Injury, poisoning and procedural complications) | 1 | 0
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 2 | 1
Urinary Urgency (Renal and urinary disorders) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1/271 | 0/127
Hypercalcemia (Investigations) | 0/271 | 1/127
Hematocrit Decreased (Investigations) | 0/271 | 1/127
Hematocrit Increased (Investigations) | 1/270 | 0/128
Hemoglobin Decreased (Investigations) | 0/270 | 1/128
Lymphocytes Decreased (Investigations) | 1/270 | 0/128
Mean Corpuscular Volume Increased (Investigations) | 1/270 | 0/128
Neutrophils Increased (Investigations) | 1/270 | 0/128
Bone Marrow Depression (Investigations) | 0/270 | 1/128

LIMITATIONS AND CAVEATS:
Efficacy endpoints are exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.